CLINICAL TRIAL: NCT07175545
Title: Enhancing Medication Adherence With Mobili®: A Crossover Randomized Controlled Trial in Portuguese Community Pharmacies
Brief Title: Testing a Smart Medication Dispenser (Mobili®) to Help People With Chronic Conditions Take Their Medicine
Acronym: MobiMAd@PT RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lusofona University (Other)
Collaborators: CBIOS - Research Center for Biosciences & Health Technologies (Unknown); MedThings (Unknown); Associação Nacional das Farmácias (Unknown); University of Oslo (Other); Universidade de Trás-os-Montes e Alto Douro (Unknown); GHTM - Global Health and Tropical Medicine (Unknown); COFAC Cooperativa de Formacao e Animacao Cultural CRL (Portugal) (Unknown)
Responsible Party: Principal Investigator, João Pedro Bernardo Gregório, PI, Universidade Lusófona de Humanidades e Tecnologias
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: LusofonaU; 2023.11968.PEX (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia)
Record Dates: First submitted 2025-08-27; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dose Administration Aids; Medication Adherence; Polypharmacy; Technology in Health; Diabetes; Cardiovascular Diseases
Keywords: Digital Health; Medication Adherence; Automatic Medicine Dispenser; Community Pharmacy
MeSH Terms: conditions — Medication Adherence; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobili® device (Intervention Group) (Experimental): Group of patients using the Mobili® device
  Interventions: Device: Independent use of the Mobili® Device by patients, overseen by pharmacists
- Placebo (Control Group) (No Intervention): Group of patients using the current Dose Administration Aid system available in the pharmacy

INTERVENTIONS:
Device: Independent use of the Mobili® Device by patients, overseen by pharmacists — After recruitment each participant will be subject to a type I medication review.
  After allocation to the intervention group, pharmacists will provide initial training to participants, and during the course of the intervention whenever necessary (e.g. when delivering the eDosette with the therapeutic regime). Pharmacists will prepare the eDosette in the pharmacy and deliver it directly to participants with no further intervention.
  Participants will receive the number of eDosettes their therapeutic regime allows, to minimize visits to the pharmacy. For the control group, pharmacists will also provide the number of DAAs the therapeutic regime allows. Upon finishing the intervention, a new type II medication review will be performed for all participants (intervention and control) and information related to their personal therapeutic regime will be provided, ensuring a safe exit of the study.
  Arms: Mobili® device (Intervention Group)

SUMMARY:
Medication adherence is one of the biggest challenges faced by healthcare systems, especially among people with multiple chronic diseases who take several medications daily. Studies show that up to half of patients do not take their medication as prescribed, which can compromise treatment effectiveness, increase complications, and lead to waste of healthcare resources.

In this context, several solutions have been developed to help patients organize their therapy, such as dose administration aids (DAAs) used in pharmacies. However, many of these systems are manual, inflexible, or difficult to use.

This study is part of the MobiMAd@PT project, which will evaluate Mobili®, a portable digital medication dispenser developed in Norway. Mobili® allows patients to automatically receive the right medication at the right time and comes with a real-time monitoring system, enabling healthcare professionals to detect missed doses and provide timely support.

The main goal of this study is to assess the effectiveness of Mobili® in improving medication adherence among patients with polypharmacy in Portugal and to understand whether this type of technology can be useful and applicable in the context of Portuguese community pharmacies. Your participation will contribute to the development of new ways to manage health at home, with the support of pharmacists and technology.

DETAILED DESCRIPTION:
Medication non-adherence is a critical challenge for global health systems, with evidence suggesting that up to half of patients may not follow their prescribed medication. Given the rates of medication non-adherence and its detrimental effects on health outcomes and health systems sustainability, numerous Dose Administration Aids (DAA) interventions have been developed. Most of them are packaging and dosage modifications, either in single and manually prepared dosette boxes, or in multidose automated dispensing (MAD) systems, prepared in community or hospital pharmacies. However, in spite of their success, most MAD are cumbersome and lack long-term sustainability.

In an era where digital health technologies are reshaping healthcare delivery, this project introduces Mobili® in Portugal, a portable MAD system developed by the Norwegian start-up Medthings. Mobili combines portability, automated dose dispensing and real-time monitoring, facilitating a more manageable medication regimen for chronic patients.

This research project aims to explore the effectiveness of Mobili on medication adherence among chronic multimorbidity patients and its adaptability in a different health system. Achieving these aims will provide valuable insights into the deployment of technology-driven interventions in actual healthcare settings, potentially transforming digital adherence solutions for chronic patients. The CFIR 2.0 Implementation Research framework will guide the development of the research tasks.

The project comprises four tasks:

1. Project management and dissemination;
2. Training of participating pharmacists, and collection of feedback on adaptability to the Portuguese context, through focus groups prior to the implementation of the intervention;
3. Assesing Mobili's efectiveness on medication adherence, through a randomized control trial (RCT) comparing Mobili users with a control group using existing DAAs;
4. developing a protocol for a future large-scale study based on tasks 2 and 3 findings.

Task 3 will also assess secondary outcomes like patient satisfaction and quality of life through interviews, using both quantitative and qualitative methods for a comprehensive intervention evaluation. The insights gained during this project will lay the groundwork for a detailed study protocol to fully assess Mobili's effectiveness in enhancing medication adherence across Europe.

This project's findings will contribute to better understand the impact of digital health interventions on medication adherence, patients' health and healthcare systems' efficiency, and will be valuable to researchers in medication adherence and implementation science. The project also holds substantial scientific and commercial potential, through:

* the deliver of a research protocol for a large-scale study to assess Mobili's clinical and economic value to European health systems
* initial insights into a disruptive DAA service business model.

The successful real-world application of the project's outcomes could enhance medication adherence and patient management, promoting a culture of adherence within the community, significantly improving care quality and generating economic benefits for patients and health systems.

The project's success strategy centers on three pillars:

1. leveraging the diverse expertise and experience within the team, with a strong support and commitment from the manufacturer of Mobili;
2. integrating Design Science with participatory action research to enhance stakeholder engagement;
3. establishing a core management team to enable a strong collaboration between scientific and clinical expertise, through regular project meetings.

The multidisciplinary research team, comprising experts in pharmaceutical services innovation, information system research, health communication, and organizational development, brings a wealth of experience from previous studies in pharmacy services, healthcare management, and digital medication adherence tools.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and above
* Non-institutionalized diabetes and cardiovascular disease patients
* At least two medications in the therapeutic regimen
* Requiring only regular oral medication that can be dispensed in the eDosette
* Able to handle the use of technological devices (i.e. smartphones)

Exclusion Criteria:

* Cognitive impairments preventing independent use of Mobili®
* Patients using medicines that do not fit or are incompatible with being dispensed in the eDosette (i.e. some capsules, solutions, insulins or GLP-1 analogues, transdermal patches, eye-drops)
* One participant per household

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Significant differences in medication adherence rates between the two groups (Objective) | From recruitment to around 6 months after
  Medication adherence rates will be measured objectively by the Pill count method, analysing how many pills are taken or forgotten by the participants
Significant differences in medication adherence rates between the two groups (Subjective) | From recruitment to around 6 months after
  Medication adherence rates will be measured subjectively by a validated medication adherence scale, using tools such as the Medical Adherence Questionnaire (MAQ) - a self-reporting instruments to measure how well patients follow their prescribed treatment regimens. Instruments like these help identify barriers to adherence, assessing adherence levels (low, medium, high).
Significant differences in medication adherence rates between the two groups (Clinical markers) | From recruitment to around 6 months after
  Monitoring clinical markers that indicate whether a medication is likely being taken, such as glycemic and arterial pressure levels, will provide additional information on adherence.

SECONDARY OUTCOMES:
Enhanced patient satisfaction, reduced incidence of medication errors, and improved quality of life measures in the intervention group | From recruitment until around 6 months after
  Patient satisfaction and quality of life measures will be measured through structured interviews with participants (both pharmacists and patients) at the start and at the end of the intervention. It is expected to use instruments such as the EuroQol Five-Dimension Questionnaire (EQ-5D) - system measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression - and similar.
Influence on the pharmacy's workflow | From recruitment until 6 months after
  There will also be a focus group with the participant pharmacists to collect additional information regarding the service integration into the pharmacy workflow.

CONTACTS AND LOCATIONS:
Overall Officials: João Pedro B Gregório, PharmD PhD, Principal Investigator — COFAC - Cooperativa Cooperativa de Animação e Formação Cultural, C.R.L
Locations (1):
- Universidade Lusófona - Centro Universitário de Lisboa, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality issues, the sharing of patient data will always be subject to request

REFERENCES:
- See also: Project Website — https://mobimadpt.wixsite.com/2025

DOCUMENTS (1):
  • Study Protocol (2025-08-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT07175545/Prot_000.pdf